CLINICAL TRIAL: NCT02189941
Title: Pilot Study of the Pharmacokinetic Profile of a Single Dose of Deferiprone Sustained-Release Formulation in Healthy Volunteers
Brief Title: Pilot Study of the Pharmacokinetic Profile of Deferiprone Sustained-Release Formulation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LA43-0114
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Deferiprone; Deferiprone sustained-release tablets; Pharmacokinetics
MeSH Terms: interventions — Deferiprone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Deferiprone sustained-release (fed) (Experimental): A single 1000 mg dose of deferiprone sustained-release following a high fat high calorie breakfast.
  Interventions: Drug: Deferiprone sustained-release
- Deferiprone sustained-release (fasting) (Experimental): A single 1000 mg dose of deferiprone sustained-release under fasting conditions.
  Interventions: Drug: Deferiprone sustained-release
- Deferiprone immediate-release (fasting) (Active Comparator): A single 1000 mg dose of Deferiprone immediate-release under fasting conditions.
  Interventions: Drug: Deferiprone immediate-release

INTERVENTIONS:
Drug: Deferiprone sustained-release — Deferiprone sustained-release tablets
  Other Names: Deferiprone
  Arms: Deferiprone sustained-release (fasting); Deferiprone sustained-release (fed)
Drug: Deferiprone immediate-release — Deferiprone immediate-release tablets
  Other Names: Ferriprox
  Arms: Deferiprone immediate-release (fasting)

SUMMARY:
The purpose of this study was to evaluate the pharmacokinetic and safety profile of the sustained-release formulation of deferiprone under both fasting and fed conditions, and evaluate the relative bioavailability of this sustained-release formulation when compared to immediate-release formulation of deferiprone under fasting conditions.

DETAILED DESCRIPTION:
This was an open-label, single-dose, randomized, three-way crossover study under fed and fasting conditions designed to determine the pharmacokinetics, safety, and tolerability of deferiprone sustained-release tablets in healthy volunteers. Subjects were randomized to receive the following 3 treatments in different orders, with a washout period of 7 days between treatments:

* 2000 mg of deferiprone sustained-release tablets under fed conditions
* 2000 mg of deferiprone sustained-release tablets under fasted conditions
* 2000 mg of Ferriprox immediate-release tablets under fasted conditions

In each period, blood samples for pharmacokinetics (PK) assessment were collected prior to dosing and at specified time points up to 24 hours post-dose. Safety assessments were conducted throughout the study.

ELIGIBILITY:
Main Inclusion Criteria:

* Meeting the age, body mass index (BMI) and weight requirements.
* Signing the Informed Consent Form.
* Acceptable alcohol and/or drug screen at check-in of each period.
* Acceptable health, blood pressure, pulse rate and temperature at check-in.
* Being a non-smoker.
* Female subjects of childbearing potential should be either sexually inactive (abstinent) for 60 days prior to the first dose of the study and throughout the study, and for 30 days after completion of the study, or be using an acceptable method of birth control.

Exclusion Criteria:

* A history of presence of significant asthma, chronic bronchitis, seizure, diabetes, migraine, hypertension, cardiovascular, pulmonary, neurological conditions, psychiatric conditions, hepatic, renal, hematopoietic or gastrointestinal diseases or ongoing infectious diseases, or any other significant abnormality as evidenced by a medical history and physical examination.
* Blood chemistry, hematology, international normalized ratio, partial thromboplastin time and urinalysis values outside clinically acceptable limits.
* A positive screen for Hepatitis B surface antigens, Hepatitis C antibodies or HIV.
* Significant abnormality found on ECG.
* Known sensitivity to deferiprone or any components of the Ferriprox tablets.
* Requiring other medication at the time of the study. Oral, injectable or topical contraceptives, and contraceptive implants are permitted as they are acceptable methods of contraception.
* Acetaminophen use within 2 weeks prior to dosing and for the duration of the study.
* History of drug or alcohol abuse within the last 6 months.
* Any known enzyme inducing or inhibiting drug taken within 30 days before the study.
* History of long QT syndrome, cardiac arrhythmias.
* Infection within two weeks prior to dosing.
* Participation in an investigational drug study within 30 days prior to first dosing in this study.
* Blood donation of 50 mL to 499 mL of whole blood within 30 days, or more than 499 mL of whole blood within 56 days prior to drug administration.
* Positive test for pregnancy at medical screening or prior to dosing in either period.
* Female subjects who are breast-feeding.
* Absolute neutrophil count (ANC) <= 1.0 x 10E9 cells/L prior to dosing for each period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gurinder Rai, MD, Principal Investigator — Apotex Inc.
Locations (1):
- Apotex Inc. BioClinical Development, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were dosed at the clinic between May and June of 2014
Pre-assignment Details: Subjects were randomized to receive 3 single-dose treatments in different sequences, with a washout of 7 days between doses. Twenty (20) subjects were screened and 12 were randomized. One subject experienced a medical event prior to the first dosing and was excluded from the study, so only 11 subjects received at least 1 dose of study product.
Groups:
- DFP-SR Fed, Then DFP-SR Fasting, Then Ferriprox Fasting: Subjects received 3 treatments in the following order, with a 7-day washout period between treatments:
  1. One dose of deferiprone sustained-release (DFP-SR) tablets under fed conditions
  2. One dose of deferiprone sustained-release tablets under fasting conditions
  3. One dose of Ferriprox immediate-release (IR) tablets under fasting conditions
- DFP-SR Fasting, Then Ferriprox Fasting, Then DFP-SR Fed: Subjects received 3 treatments in the following order, with a 7-day washout period between treatments:
  1. One dose of deferiprone sustained-release tablets under fasting conditions
  2. One dose of Ferriprox immediate-release tablets under fasting conditions
  3. One dose of deferiprone sustained-release tablets under fed conditions
- Ferriprox Fasting, Then DFP-SR Fed, Then DFP-SR Fasting: Subjects received 3 treatments in the following order, with a 7-day washout period between treatments:
  1. One dose of Ferriprox immediate-release tablets under fasting conditions
  2. One dose of deferiprone sustained-release tablets under fed conditions
  3. One dose of deferiprone sustained-release tablets under fasting conditions
Period: Overall Study
Arm/Group | DFP-SR Fed, Then DFP-SR Fasting, Then Ferriprox Fasting | DFP-SR Fasting, Then Ferriprox Fasting, Then DFP-SR Fed | Ferriprox Fasting, Then DFP-SR Fed, Then DFP-SR Fasting
Started | 4 | 4 | 3
Completed | 4 | 4 | 2
Not Completed | 0 | 0 | 1
Not completed — Non-compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteers: Subjects received one dose of deferiprone sustained-release tablets under fed conditions, one dose of deferiprone sustained-release tablets under fasting conditions, and one dose of deferiprone immediate-release tablets under fasting conditions, 7 days apart
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 3
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 11

OUTCOME MEASURES:

1. Primary Outcome: AUCt for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: AUCt (Area Under the Curve to the last measured time) was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite. Blood samples were obtained prior to dosing and at 0.25, 0.5, 0.75, 1, 1.3333, 1.6667, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16 and 24 hours post-dose.
Time Frame: 24-hour interval
Population: All subjects who contributed evaluable pharmacokinetics data
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Groups:
- Deferiprone Sustained-release (Fed): A single 2000 mg dose of deferiprone sustained-release following a high fat high calorie breakfast.
  Deferiprone sustained-release: Deferiprone sustained-release tablets
- Deferiprone Sustained-release (Fasting): A single 2000 mg dose of deferiprone sustained-release under fasting conditions.
  Deferiprone sustained-release: Deferiprone sustained-release tablets
- Deferiprone Immediate-release (Fasting): A single 2000 mg dose of Deferiprone immediate-release under fasting conditions.
  Deferiprone immediate-release: Deferiprone immediate-release tablets
Arm/Group | Deferiprone Sustained-release (Fed) | Deferiprone Sustained-release (Fasting) | Deferiprone Immediate-release (Fasting)
Number analyzed (Participants) | 10 | 10 | 11
mcg*h/mL
  Deferiprone | 63.5 (10.0) | 52.3 (14.8) | 71.1 (10.9)
  Deferiprone 3-O-glucuronide | 171.9 (33.4) | 147.2 (41.5) | 192.7 (32.8)

2. Primary Outcome: AUCinf for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: AUCinf (Area Under the Curve to infinity) was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite. Blood samples were obtained prior to dosing and at 0.25, 0.5, 0.75, 1, 1.3333, 1.6667, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16 and 24 hours post-dose.
Time Frame: 24-hour interval
Population: All subjects who contributed evaluable pharmacokinetics data
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Deferiprone Sustained-release (Fed) | Deferiprone Sustained-release (Fasting) | Deferiprone Immediate-release (Fasting)
Number analyzed (Participants) | 10 | 10 | 11
mcg*h/mL
  Deferiprone | 66.2 (11.1) | 57.2 (16.1) | 71.6 (11.0)
  Deferiprone 3-O-glucuronide | 181.3 (39.9) | 169.2 (62.3) | 193.4 (32.5)

3. Primary Outcome: Cmax for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Cmax (maximum concentration in the serum) was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite. Blood samples were obtained prior to dosing and at 0.25, 0.5, 0.75, 1, 1.3333, 1.6667, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16 and 24 hours post-dose.
Time Frame: 24-hour interval
Population: All subjects who contributed evaluable pharmacokinetics data
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Deferiprone Sustained-release (Fed) | Deferiprone Sustained-release (Fasting) | Deferiprone Immediate-release (Fasting)
Number analyzed (Participants) | 10 | 10 | 11
mcg/mL
  Deferiprone | 8.7 (1.8) | 5.8 (1.6) | 21.9 (6.9)
  Deferiprone 3-O-glucuronide | 18.5 (4.2) | 14.3 (2.9) | 33.2 (5.0)

4. Primary Outcome: Tmax for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Tmax (the time to Cmax) was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite. Blood samples were obtained prior to dosing and at 0.25, 0.5, 0.75, 1, 1.3333, 1.6667, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16 and 24 hours post-dose.
Time Frame: 24-hour interval
Population: All subjects who contributed evaluable pharmacokinetics data
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Deferiprone Sustained-release (Fed) | Deferiprone Sustained-release (Fasting) | Deferiprone Immediate-release (Fasting)
Number analyzed (Participants) | 10 | 10 | 10
h
  Deferiprone | 4.4 (0.9) | 3.3 (1.4) | 1.3 (1.1)
  Deferiprone 3-O-glucuronide | 6.0 (1.5) | 4.5 (1.5) | 3.0 (0.9)

5. Primary Outcome: Thalf for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Thalf (the apparent terminal elimination half-life of the drug) was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite. Blood samples were obtained prior to dosing and at 0.25, 0.5, 0.75, 1, 1.3333, 1.6667, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16 and 24 hours post-dose.
Time Frame: 24-hour interval
Population: All subjects who contributed evaluable pharmacokinetics data
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Deferiprone Sustained-release (Fed) | Deferiprone Sustained-release (Fasting) | Deferiprone Immediate-release (Fasting)
Number analyzed (Participants) | 10 | 10 | 11
h
  Deferiprone | 2.8 (1.4) | 5.0 (3.5) | 1.9 (0.3)
  Deferiprone 3-O-glucuronide | 3.7 (3.4) | 6.1 (4.9) | 2.4 (0.5)

6. Secondary Outcome: Safety and Tolerability of Deferiprone Sustained Release Tablets
Description: The number of participants who experienced adverse events between the time of dosing up to 24 hours post-dose, including any changes of clinical significance in vital signs, 12-lead ECG, and clinical laboratory tests
Time Frame: From time of dose until 24 hours post dose
Population: All subjects who received at least one dose of study medication and had at least one safety assessment
Measure: Number; unit: participants
Arm/Group | Deferiprone Sustained-release (Fed) | Deferiprone Sustained-release (Fasting) | Deferiprone Immediate-release (Fasting)
Number analyzed (Participants) | 10 | 10 | 11
participants | 5 | 5 | 6

ADVERSE EVENTS:
Time Frame: 1 day
Description: Safety data were collected from the time of dosing up to 24 hours post-dose
Arm/Group | Deferiprone Sustained-release (Fed) | Deferiprone Sustained-release (Fasting) | Deferiprone Immediate-release (Fasting)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 5/10 | 5/10 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferiprone Sustained-release (Fed) (N=10) | Deferiprone Sustained-release (Fasting) (N=10) | Deferiprone Immediate-release (Fasting) (N=11)
Heart rate decreased (Investigations) | 2 (3) | 2 (2) | 2 (3)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Catheter site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes